CLINICAL TRIAL: NCT06110494
Title: A New Clinical Use of Ferumoxytol Nanoparticles: An Antibiofilm Treatment
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Principal Investigator, Bekir Karabucak, Chair of The Endodontics Department, University of Pennsylvania
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 828211
Record Dates: First submitted 2023-10-25; First posted 2023-10-31 (Actual); Results first posted 2024-08-28 (Actual); Last update posted 2024-08-28 (Actual); Status verified 2024-08

CONDITIONS: Apical Periodontitis; Pulp Disease, Dental
Keywords: Pulp infection; Nanotechnology; antibacterial; disinfection; iron oxide nanoparticles
MeSH Terms: conditions — Periapical Periodontitis; Dental Pulp Diseases | interventions — Iron, Dietary; Ferrosoferric Oxide; Sodium Hypochlorite; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Iron oxide nanoparticles treatment Ferumoxytol/H2O2 (Experimental): After access preparation with sterile burs and sterile saline irrigation and working length determination as part of routine root canal treatment, and after obtaining a pre-treatment bacteriological samples, 2 mL of a mixture of Ferumoxytol (6mg/mL)/H2O2(3%) was introduced into the canal. Canals were instrumented with 15/0.04, 20/0.04, and 25/0.04 rotary files using 2 mL of treatment solution after each file with a total of 8 mL of solution used and a total contact time of 10 minutes.
  Interventions: Drug: Iron oxide nanoparticles treatment Ferumoxytol/H2O2; Drug: supplementary irrigation
- Sodium Hypochlorite (NaOCl) (Active Comparator): After access preparation with sterile burs and sterile saline irrigation and working length determination as part of routine root canal treatment, and after obtaining a pre-treatment bacteriological samples, 2 mL of 3% NaOCl was introduced into the canal. Canals were instrumented with 15/0.04, 20/0.04, and 25/0.04 rotary files using 2 mL of solution after each file with a total of 8 mL of treatment solution used and a total contact time of 10 minutes.
  Interventions: Drug: NaOCl; Drug: supplementary irrigation
- Saline (NaCl) (Placebo Comparator): After access preparation with sterile burs and sterile saline irrigation and working length determination as part of routine root canal treatment, and after obtaining a pre-treatment bacteriological samples, 2 mL of 0.89% NaCl was introduced into the canal. Canals were instrumented with 15/0.04, 20/0.04, and 25/0.04 rotary files using 2 mL of treatment solution after each file with a total of 8 mL of solution used and a total contact time of 10 minutes.
  Interventions: Drug: NaCl; Drug: supplementary irrigation

INTERVENTIONS:
Drug: Iron oxide nanoparticles treatment Ferumoxytol/H2O2 — Participants receive a topical treatment through a root canal irrigation needle containing A mixture of 6mg/mL Ferumoxytol nanoparticles solution mixed with 3% H2O2 for 10 minutes contact time
  Other Names: Fer; Feraheme
  Arms: Iron oxide nanoparticles treatment Ferumoxytol/H2O2
Drug: NaOCl — Participants receive a topical treatment through a root canal irrigation needle containing 3% NaOCl for 10 minutes contact time
  Other Names: Sodium Hypochlorite; Active comparator
  Arms: Sodium Hypochlorite (NaOCl)
Drug: NaCl — Participants receive a topical treatment through a root canal irrigation needle containing 0.89% NaCl for 10 minutes contact time
  Other Names: Placebo comparator; saline
  Arms: Saline (NaCl)
Drug: supplementary irrigation — All canals in all groups were irrigated with 2 mL of 3% NaOCl, followed by ultrasonic irrigant activation for 30s twice.
  seconds. This step was repeated once again making the total activation time 1 min and the total contact time of the irrigant 3 min. Upon completion of irrigation, a third bacterial sample (S3) was taken following the deactivation, washing, drying, and sampling steps as described previously
  Other Names: NaOCl with passive ultrasonic activation; adjunctive irrigation step

SUMMARY:
The goal of this observational is study is to develop a protocol for root canal biofilms disinfection using a clinically approved and commercially available iron oxide nanoparticle formulation Ferumoxytol/H2O2 treatments. This protocol will be testing local single topical application of Ferumoxytol within the root canal system in patients going through routine root canal treatment, evaluate its potential as anti-biofilm treatment and compare it to the clinical gold standard disinfecting solution sodium hypochlorite (positive control) and saline (negative control).

DETAILED DESCRIPTION:
Patients presenting to the Department of Endodontics, School of Dental Medicine, University of Pennsylvania for evaluation and routine endodontic treatment of infected, necrotic teeth with chronic apical periodontitis will be asked to take part in the study if they meet the inclusion criteria and volunteer to participate. After eligibility of the patient is confirmed, the patient will be assigned to treatments through the process of drawing lots from a box that was maintained in a locked cabinet. Before treatment, patients will be thoroughly informed about the nature, potential risks and alternatives of the study as well as the root canal treatment. Patients will be presented with a written consent form regarding the above mentioned study characteristics as well as the regular consent forms for the root canal therapy, including the consent form for endodontic treatement, acknowledgement of privacy practices and a patient understanding and informed consent form. Briefly, the patient will be anesthetized and the tooth isolated with rubber dam. 30% H2O2 followed by 3% NaOCl will be used to disinfect the tooth and the rubber dam. The removal of caries and the endodontic access will be carried out by sterile high-speed carbide burs.After access preparation with sterile burs and sterile saline irrigation, thermoplastic gutta percha was placed to temporarily block the orifice. The field, including the pulp chamber, is cleaned and disinfected as described previously. NaOCl is neutralized with 10% sodium thiosulfate. Contamination control sample (S0) will be taken from the internal cavosurface angle where the paper points will accidentally touch during sampling.After initial access to the root canal orifices, working length will be measured and a bacteriological sample will be taken from the targeted canals (S1). Sterile paper points will be placed into the canal, allowed to saturate and then transferred to a vial containing liquid dental transport media (LDT). For NaOCl group (Positive control), canals will be instrumented up to size 25/0.04 taper using 2mL of 3% NaOCl in between files. For Ferumoxytol/H2O2 group, canals will be instrumented up to size 25/0.04 taper using 2mL of a mixture of 6 mg/ml of Ferumoxytol with 3% H2O2. For saline only group, canals will be instrumented up to size 25/0.04 taper using 2mL of saline. When the final 25/0.04 taper apical size is reached, a second bacterial sample will be taken (S2). Before all samplings, sodium hypochlorite, Feramehe/ H2O2 and Saline. Canal contents will be deactivated with sodium thiosulphate for NaOCl,and saline wash will be used for Fer/H2O2 and saline treatments. A wash step with 1 mL saline was done to wash the deactivating solution, and paper points were used to dry the canals. A second bacterial sample was taken (S2) by placing LDT inside the canal, agitating it with 25/0.02 Hedstrom hand file, followed by absorbing the content with 2 paper points placed in the canal for 30 seconds each. The paper points will be placed inside a tube containing LDT. An additional step was included for all the test groups to evaluate if further irrigation after (S2) will lead to more reduction of bacterial counts inside the root canal system. This could inform future experiments evaluating the possibility of synergistic antimicrobial effects for the sequential Fer/H2O2 and NaOCl treatment. All canals in all groups were irrigated with 2 mL of 3% NaOCl (1 min), followed by ultrasonic irrigant activation for 30 seconds. This step was repeated once again making the total activation time 1 min and the total contact time of the irrigant 3 min. Upon completion of irrigation, a third bacterial sample (S3) was taken following the deactivation, washing, drying, and sampling steps as described previously. The remaining treatment sequences of the routine root canal therapy will be carried out after these procedures including further root-end enlargement and final routine irrigation protocol. The root canals will be dried with paper points, a medication (calcium hydroxide) will be placed and the teeth sealed with a temporary restoration. Patients will return after one to four weeks for completion of the root filling. For the any of the groups, the treatment procedures carried out during this investigation do not differ from the standard root canal treatment protocol with the exception of additional irrigation step with the experimental solution and the bacteriologic sampling procedures. The paper points used to take the bacteriological sampling will be transferred to the microbiology laboratory using a vial containing 1 ml of LDT. The laboratory procedures will be performed at the University of Pennsylvania Leon Levy Oral Health Sciences Building of the School of Dental Medicine in the Microbiology Laboratory Vial labels will contain information on tooth number, sample number (S0-S1-S2-S3) and the experimental group. The samples will be diluted and plated in culture plates. The culture plates will be incubated at 37°C in an anaerobic glove box containing 5% hydrogen, 5% CO2 and balance N2 for 5 days. After incubation the number of colony forming units will be determined by using a stereoscope. ANOVA and Students t-test will be used for statistical analysis.

ELIGIBILITY:
Inclusion Criteria:

1. Patients to welling to participate in the study.
2. Patients are 18 years or above.
3. Non-contributory medical history (Patient can be seen for regular dental appointment in PDM; ASA classes I and II).
4. Tooth requiring root canal treatment with radiographic presence of periapical radiolucency and responding to thermal sensitivity testing negatively (difluordichlormethane at 50 °C) (Endo-Ice, Coltène/Whaledent Inc., Cuyahoga Falls, Ohio) and Negatively to EPT testing.
5. Tooth with adequate remaining tooth structure for proper isolation with rubber dam.
6. No history of previous endodontic treatment on the tooth.
7. Teeth with single canal and single and roots with single canals in multirooted teeth.

Exclusion Criteria:

1. Self-reported Pregnancy.
2. Patients requiring antibiotic premedication prior to dental treatment.
3. Patients with multiple drug allergies.
4. Patients with known hypersensitivity to Ferumoxytol nanoparticles or any iron products.
5. Patients who are scheduled for MRI for the head region within three months after Fer nanoparticles application.
6. Periodontal changes (pockets 3 mm, mobility Grade I or gingival edema).
7. Radiographic presence of resorptive processes.
8. Cracked and fractured teeth.
9. if one of the inclusion criteria is not met

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2020-07-13 (Actual); Primary Completion 2022-03-10 (Actual); Study Completion 2022-03-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bekir Karabucak, DMD, MS, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
Only the participants chart numbers were collected during the study. The study protocol, statistical analysis plan and informed consent form will be published as supporting information with the final manuscript
Supporting Information: Study Protocol, SAP, ICF
Time Frame: the supporting information will be available with the publication

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients presenting to the Department of Endodontics, School of Dental Medicine, University of Pennsylvania for evaluation and routine endodontic treatment of infected, necrotic teeth with chronic apical periodontitis were asked if they would like to take part in the study and volunteer to participate.
Pre-assignment Details: Forty-four (44) patients presenting to the endodontic with an initial diagnosis of pulp necrosis were assessed for eligibility. Seven (7) patients were initially excluded during the eligibility assessment (not meeting inclusion criteria (n=4);declined to participate (n=3). five patients were part of a pilot to test different bacterial sampling methods prior to the experimental phase
Units Other Than Participants: roots
Period: Overall Study
Arm/Group | Iron Oxide Nanoparticles Treatment Ferumoxytol/H2O2 | Sodium Hypochlorite (NaOCl) | Saline (NaCl)
Started | 11; 11 roots | 11; 11 roots | 10; 10 roots
Completed | 8; 8 roots | 10; 10 roots | 9; 9 roots
Not Completed | 3; 3 roots | 1; 1 roots | 1; 1 roots
Not completed — Protocol Violation | 2 | 0 | 1
Not completed — Dixon's test for outlier analysis | 1 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Iron Oxide Nanoparticles Treatment Ferumoxytol/H2O2 | Sodium Hypochlorite (NaOCl) | Saline (NaCl) | Total
Number analyzed (Participants) | 11 | 11 | 10 | 32
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 11 | 11 | 10 | 32
  Between 18 and 65 years | 0 | 0 | 0 | 0
  >=65 years | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Sex of the participants was not collected as baseline information during the study
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 11 | 11 | 10 | 32

OUTCOME MEASURES:

1. Primary Outcome: The Primary Outcome Parameter Will be the Difference in Bacterial Reduction Between the Experimental and Control Disinfection Groups Group (Ferumoxytol) and Comparison Groups (Positive and Negative Controls).
Description: This study is designed to evaluate the antibacterial efficacy of Ferumoxytol/H2O2 and to compare it to the gold standard disinfection solution (NaOCl) and negative control solution (NaCl). The outcome will be evaluated by taking bacterial samples from the root canals during routine root canal treatment before and after applying different disinfection protocols. The disinfection efficacy was calculated by comparing the difference in microbial CFU reduction (post treatment sample/pretreatment sample) between the three disinfection protocols
Time Frame: baseline (pretreatment) and after 10 minutes of treatment (post treatment)
Population: The antimicrobial effectiveness of Fer/H2O2 was evaluated by calculating the CFU log reduction of the viable microbial counts between pretreatment sample S1 and the post treatment sample S2 and compare it with the CFU log reduction of NaOCL and NaCl
Measure: Median (Inter-Quartile Range); unit: CFU log reduction
Units Other Than Participants: Roots
Arm/Group | Iron Oxide Nanoparticles Treatment Ferumoxytol/H2O2 | Sodium Hypochlorite (NaOCl) | Saline (NaCl)
Number analyzed (Participants) | 7 | 10 | 9
Number analyzed (Roots) | 7 | 10 | 9
CFU log reduction | 0.0002300 [0.0000559 to 0.001890] | 0.0001056 [0.0000146 to 0.2104] | 0.01196 [0.002769 to 0.05574]
Statistical Analysis 1: Comparison: Iron Oxide Nanoparticles Treatment Ferumoxytol/H2O2 vs Sodium Hypochlorite (NaOCl) vs Saline (NaCl); The sample size estimate was calculated in Pass Software 2021, using a test that compares the ratio of two means from independent samples using data that has been log-normalized. An alpha of 0.05 and power of 80% was assumed, with means and standard deviations pulled from previous studies that employed similar methodology. This produced a required sample size of 16 for each group. Pairwise comparisons were done using Mann-Whitney U test to compare the antimicrobial effectiveness; Test type: Other — Pairwise comparisons were done using Mann-Whitney U test of log10 transformed CFU reduction data to compare the antimicrobial effectiveness; p = 0.05, Wilcoxon (Mann-Whitney) — Pairwise comparisons were done using Mann-Whitney U test of log 10 transformed data to compare the antimicrobial effectiveness of Fer/H2O2 in comparison with the negative (saline) and positive (NaOCl) controls with P values set at < 0.05

2. Secondary Outcome: The Effect of Additional (Supplementary) Irrigation and Adjunctive Irrigant (NaOCl) Activation Using Passive Ultrasonic Activation After Irrigation With Experimental and Control Irrigants.
Description: All groups received an additional irrigation step with NaOCl with passive ultrasonic activation. An additional step was included for all the test groups to evaluate if further irrigation after (S2) will lead to more reduction of bacterial counts inside the root canal system. This could inform future experiments evaluating the possibility of synergistic antimicrobial effects for the sequential ferumoxytol and NaOCl treatment.
Time Frame: the baseline of this measurement starts right after treatment with either experimental, negative or positive control agent (S2). This measurement ends after irrigating the canals with NaOCl and irritant activation for 3 minutes.
Population: The antimicrobial effectiveness of supplementary irrigation was evaluated by calculating the CFU log reduction of the viable microbial counts between post treatment sample S2 and the post supplementary irrigation sample S3 and compare it with the CFU log reduction of NaOCL and NaCl (positive and negative controls)
Measure: Median (Inter-Quartile Range); unit: CFU log reduction
Units Other Than Participants: roots
Groups:
- Iron Oxide Nanoparticles Treatment Ferumoxytol/H2O2: After access preparation with sterile burs and sterile saline irrigation and working length determination as part of routine root canal treatment, and after obtaining a pre-treatment bacteriological samples, 2 mL of a mixture of Ferumoxytol (6mg/mL)/H2O2(3%) was introduced into the canal. Canals were instrumented with 15/0.04, 20/0.04, and 25/0.04 rotary files using 2 mL of treatment solution after each file with a total of 8 mL of solution used and a total contact time of 10 minutes.
  Iron oxide nanoparticles treatment Ferumoxytol/H2O2: Participants receive a topical treatment through a root canal irrigation needle containing A mixture of 6mg/mL Ferumoxytol nanoparticles solution mixed with 3% H2O2 for 10 minutes contact time
  supplementary irrigation: All canals in all groups were irrigated with 2 mL of 3% NaOCl, followed by ultrasonic irrigant activation for 30s twice.
  seconds. This step was repeated once again making the total activation time 1 min and the total contact time of the irrigant 3 min. Upon completion of irrigation, a third bacterial sample (S3) was taken following the deactivation, washing, drying, and sampling steps as described previously
- Sodium Hypochlorite (NaOCl): After access preparation with sterile burs and sterile saline irrigation and working length determination as part of routine root canal treatment, and after obtaining a pre-treatment bacteriological samples, 2 mL of 3% NaOCl was introduced into the canal. Canals were instrumented with 15/0.04, 20/0.04, and 25/0.04 rotary files using 2 mL of solution after each file with a total of 8 mL of treatment solution used and a total contact time of 10 minutes.
  NaOCl: Participants receive a topical treatment through a root canal irrigation needle containing 3% NaOCl for 10 minutes contact time
  supplementary irrigation: All canals in all groups were irrigated with 2 mL of 3% NaOCl, followed by ultrasonic irrigant activation for 30s twice.
  seconds. This step was repeated once again making the total activation time 1 min and the total contact time of the irrigant 3 min. Upon completion of irrigation, a third bacterial sample (S3) was taken following the deactivation, washing, drying, and sampling steps as described previously
- Saline (NaCl): After access preparation with sterile burs and sterile saline irrigation and working length determination as part of routine root canal treatment, and after obtaining a pre-treatment bacteriological samples, 2 mL of 0.89% NaCl was introduced into the canal. Canals were instrumented with 15/0.04, 20/0.04, and 25/0.04 rotary files using 2 mL of treatment solution after each file with a total of 8 mL of solution used and a total contact time of 10 minutes.
  NaCl: Participants receive a topical treatment through a root canal irrigation needle containing 0.89% NaCl for 10 minutes contact time
  supplementary irrigation: All canals in all groups were irrigated with 2 mL of 3% NaOCl, followed by ultrasonic irrigant activation for 30s twice.
  seconds. This step was repeated once again making the total activation time 1 min and the total contact time of the irrigant 3 min. Upon completion of irrigation, a third bacterial sample (S3) was taken following the deactivation, washing, drying, and sampling steps as described previously
Arm/Group | Iron Oxide Nanoparticles Treatment Ferumoxytol/H2O2 | Sodium Hypochlorite (NaOCl) | Saline (NaCl)
Number analyzed (Participants) | 8 | 9 | 9
Number analyzed (roots) | 8 | 9 | 9
CFU log reduction | 1.000 [0.4345 to 2.453] | 1 [0.1472 to 6.000] | 0.1360 [0.02710 to 8.400]

3. Secondary Outcome: The Overall Effect of Antimicrobial Irrigation of Infected Root Canals Using Experimental and Control Irrigants, in Addition to Supplementary Irrigant (NaOCl) Activation.
Description: All groups received treated with either Experimental (ferumoxytol), NaOCl (positive control) or Saline (NaCl, negative control). Followed by supplementary irrigation and activation. This could inform future experiments evaluating the possibility of synergistic antimicrobial effects for the sequential ferumoxytol and NaOCl treatment.
Time Frame: This measure starts at baseline (pretreatment) (S1). This measure ends after 10 minutes of treatment with either experimental, positive or negative control irrigants and additional 3 minutes of supplementary irrigation (S3)
Population: The overall antimicrobial effectiveness of antimicrobial irrigation was evaluated by calculating the CFU log reduction of the viable microbial counts between baseline pretreatment sample (S1) and the post supplementary irrigation sample (S3). The CFU log reduction was compared between the groups (experimental and controls)
Measure: Median (Inter-Quartile Range); unit: CFU log reduction
Units Other Than Participants: roots
Arm/Group | Iron Oxide Nanoparticles Treatment Ferumoxytol/H2O2 | Sodium Hypochlorite (NaOCl) | Saline (NaCl)
Number analyzed (Participants) | 7 | 9 | 9
Number analyzed (roots) | 7 | 9 | 9
CFU log reduction | 0.0002360 [0.0001580 to 0.001890] | 0.0001590 [0.00004078 to 0.05725] | 0.001630 [0.0002660 to 0.05380]

ADVERSE EVENTS:
Time Frame: The participation of the participants in this study was within the time necessary for the standard routine single visit root canal therapy. Monitoring of blood pressure and signs and symptoms of hypersensitivity during the next 30 minutes after Ferumoxytol application, during which the remaining treatment sequences of the routine root canal therapy will be carried out. After the procedure was done, the study relied on self reporting by the participant by a routine post-op call the next day.
Description: There are no potential risks associated with noninvasive bacteriological sampling. Ferumoxytol with much higher concentrations has been FDA approved and used in medicine as IV to treat iron deficiency anemia. Ferumoxytol used in this study is applied topically and is limited within the root canal system which is devoid of blood supply and was not used systemically. Exclusion criteria was set to exclude participants at risk of developing adverse events reported with systemic applications.
Arm/Group | Iron Oxide Nanoparticles Treatment Ferumoxytol/H2O2 | Sodium Hypochlorite (NaOCl) | Saline (NaCl)
All-Cause Mortality (participants affected / at risk) | 0/11 | 0/11 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/11 | 0/10
Other Adverse Events (participants affected / at risk) | 0/11 | 0/11 | 0/10

LIMITATIONS AND CAVEATS:
we emphasize the limitation of our clinical study. Limitations include the small sample size

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-12-17): https://cdn.clinicaltrials.gov/large-docs/94/NCT06110494/Prot_SAP_003.pdf
  • Informed Consent Form (2021-12-17): https://cdn.clinicaltrials.gov/large-docs/94/NCT06110494/ICF_002.pdf